CLINICAL TRIAL: NCT02305381
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Placebo as add-on to Basal Insulin Alone or Basal Insulin in Combination With Metformin in Subjects With Type 2 Diabetes
Acronym: SUSTAIN™ 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3627; 2013-004502-26 (EudraCT Number); U1111-1149-3738 (Other: WHO); JapicCTI-142729 (Other: JAPIC)
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 0.5 mg/Week (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg/Week (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide Placebo 0.5 mg/Week (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide Placebo 1.0 mg/Week (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Injected subcutaneously (s.c. under the skin) once-weekly. As add-on to the pre-trial background medication.
  Arms: Semaglutide 0.5 mg/Week; Semaglutide 1.0 mg/Week
Drug: placebo — Injected subcutaneously (s.c. under the skin) once-weekly. As add-on to the pre-trial background medication.
  Arms: Semaglutide Placebo 0.5 mg/Week; Semaglutide Placebo 1.0 mg/Week

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of the trial is to investigate efficacy and safety of semaglutide once weekly versus placebo as add-on to basal insulin alone or basal insulin in combination with metformin in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age at least 18 years at the time of signing inform consent. For Japan: Male or female, age at least 20 years at the time of signing informed consent - Subjects diagnosed with T2DM (type 2 diabetes mellitus) and on stable diabetes treatment (plus/minus 20 percent change in total daily dose) with basal insulin (minimum of 0.25 IU/kg/day and/or 20 IU/day of: insulin glargine, insulin detemir, insulin degludec and/or NPH insulin) alone or in combination with metformin (minimum of 1500 mg/day or maximal tolerable dose) for 90 days prior to screening - HbA1c (glycosylated haemoglobin) 7.0 - 10.0 percent (53 - 86 mmol/mol) both inclusive Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method throughout the trial including the 5 weeks follow-up period (adequate contraceptive measures as required by local regulation or practice). Germany: Only highly effective methods of birth control are accepted (ie one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine device), or sexual abstinence or vasectomised partner. Japan: Adequate contraceptive measures are abstinence (not having sex), diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives - Treatment with any glucose lowering agents other than stated in the inclusion criteria in a period of 90 days before screening. An exception is short-term treatment (7 days or less in total) with bolus insulin in connection with intercurrent illness - Experienced more than 3 episodes of severe hypoglycaemia within 6 months prior to screening, and/or hypoglycaemia unawareness - History of pancreatitis (acute or chronic) - Screening calcitonin value above or equal to 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome 2 (MEN 2) - Severe renal impairment defined as eGFR (estimated glomerular filtration rate) below 30 mL/min/1.73 m^2 per Modification of Diet in Renal Disease (MDRD) formula (4 variable version) - Acute coronary or cerebrovascular event within 90 days before randomisation - Heart failure, New York Heart Association (NYHA) Class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-11-21 (Actual); Study Completion 2015-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (91):
- United States (66):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Fleming Island, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gillespie, Illinois
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Overland Park, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Yukon, Oklahoma
  - Novo Nordisk Investigational Site, Levittown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Athens, Tennessee
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Germany (10):
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
- Japan (6):
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Novi Sad
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Prešov

REFERENCES:
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Result] Rodbard H, Lingvay I, Reed J, de la Rosa R, Rose L, Sugimoto D, Araki E, Chu P-L, Wijayasinghe N, Norwood P. Efficacy and safety of semaglutide once-weekly vs placebo as add-on to basal insulin alone or in combination with metformin in subjects with type 2 diabetes (SUSTAIN 5). Diabetologia. 2016; 59: S364-5.
- [Result] Rodbard HW, Lingvay I, Reed J, de la Rosa R, Rose L, Sugimoto D, Araki E, Chu PL, Wijayasinghe N, Norwood P. Semaglutide Added to Basal Insulin in Type 2 Diabetes (SUSTAIN 5): A Randomized, Controlled Trial. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2291-2301. doi: 10.1210/jc.2018-00070. PMID 29688502
- [Result] Warren M, Chaykin L, Trachtenbarg D, Nayak G, Wijayasinghe N, Cariou B. Semaglutide as a therapeutic option for elderly patients with type 2 diabetes: Pooled analysis of the SUSTAIN 1-5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2291-2297. doi: 10.1111/dom.13331. Epub 2018 Jun 7. PMID 29687620
- [Result] Ahren B, Atkin SL, Charpentier G, Warren ML, Wilding JPH, Birch S, Holst AG, Leiter LA. Semaglutide induces weight loss in subjects with type 2 diabetes regardless of baseline BMI or gastrointestinal adverse events in the SUSTAIN 1 to 5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2210-2219. doi: 10.1111/dom.13353. Epub 2018 Jun 12. PMID 29766634
- [Result] DeVries JH, Desouza C, Bellary S, Unger J, Hansen OKH, Zacho J, Woo V. Achieving glycaemic control without weight gain, hypoglycaemia, or gastrointestinal adverse events in type 2 diabetes in the SUSTAIN clinical trial programme. Diabetes Obes Metab. 2018 Oct;20(10):2426-2434. doi: 10.1111/dom.13396. Epub 2018 Jul 9. PMID 29862621
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Jendle J, Birkenfeld AL, Polonsky WH, Silver R, Uusinarkaus K, Hansen T, Hakan-Bloch J, Tadayon S, Davies MJ. Improved treatment satisfaction in patients with type 2 diabetes treated with once-weekly semaglutide in the SUSTAIN trials. Diabetes Obes Metab. 2019 Oct;21(10):2315-2326. doi: 10.1111/dom.13816. Epub 2019 Jul 12. PMID 31215727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 90 sites in 5 countries, as follows: Germany: 10 sites; Japan: 6 sites; Serbia: 4 sites; Slovakia: 5 sites; United States: 65.
Groups:
- Semaglutide 0.5 mg: Subjects received semaglutide 0.25 mg subcutaneous (sc) injection once weekly for 4 weeks followed by semaglutide 0.5 mg once weekly up to week 30. Semaglutide injection was administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same day of the week during the trial.
- Semaglutide 1.0 mg: Subjects received semaglutide 0.25 mg sc injection once weekly for 4 weeks followed by semaglutide 0.5 mg once weekly for next 4 weeks and then semaglutide 1.0 mg once weekly up to week 30.Semaglutide injection was administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same day of the week during the trial.
- Placebo: Subjects received placebo (matched to semaglutide) sc injection once weekly for 30 weeks. Placebo injection was administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same day of the week during the trial.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Started | 132 | 132 | 133
Exposed | 132 | 131 | 133
Premature Discontinuation of Treatment | 14 (Subjects who prematurely discontinued treatment were allowed to continue participation in the trial.) | 16 (Subjects who prematurely discontinued treatment were allowed to continue participation in the trial) | 13 (Subjects who prematurely discontinued treatment were allowed to continue participation in the trial.)
Completed | 127 (Subjects who completed the trial.) | 127 (Subjects who completed the trial.) | 126 (Subjects who completed the trial.)
Not Completed | 5 | 5 | 7
Not completed — Unclassified | 5 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set which included all randomised subjects who had received at least 1 dose of randomised semaglutide or placebo.
Groups:
- Semaglutide 0.5 mg: Subjects received semaglutide 0.25 mg sc injection once weekly for 4 weeks followed by semaglutide 0.5 mg once weekly up to week 30. Semaglutide injection was administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same day of the week during the trial.
- Semaglutide 1.0 mg: Subjects received semaglutide 0.25 mg sc injection once weekly for 4 weeks followed by semaglutide 0.5 mg once weekly for next 4 weeks and then semaglutide 1.0 mg once weekly up to week 30. Semaglutide injection was administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same day of the week during the trial.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo | Total
Number analyzed (Participants) | 132 | 131 | 133 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.3) | 58.5 (9.0) | 58.8 (10.9) | 58.8 (10.1)
Age, Customized [Number; unit: participants]
  Adults (18-64 years) | 93 | 102 | 86 | 281
  From 65-84 years | 39 | 29 | 46 | 114
  85 years and over | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 54 | 62 | 174
  Male | 74 | 77 | 71 | 222
Glycosylated haemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.36 (0.83) | 8.31 (0.82) | 8.42 (0.88) | 8.37 (0.84)
Body weight [Mean (Standard Deviation); unit: kg] | 92.74 (19.57) | 92.49 (22.23) | 89.88 (21.06) | 91.70 (20.97)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 161.0 (62.38) | 152.5 (50.91) | 154.1 (46.66) | 155.9 (53.68)
Insulin dose [Median (Full Range); unit: international unit] — Population: Number of participants analysed=participants with available data for insulin dose at baseline.
  international unit
    number analyzed (Participants) | 131 | 131 | 133 | 395
    (all) | 35.00 [15.00 to 300.00] | 36.00 [14.00 to 320.00] | 36.00 [12.00 to 124.00] | 36.00 [12.00 to 320.00]
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 78.89 (9.72) | 78.73 (9.98) | 79.35 (9.71) | 78.99 (9.79)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 134.87 (15.00) | 134.40 (16.32) | 134.99 (16.68) | 134.76 (15.98)
Diabetes Treatment Satisfaction Questionnaire [Mean (Standard Deviation); unit: scores on scale] — The DTSQs questionnaire was used to assess subjects' treatment satisfaction and contained 8 components and evaluates the diabetes treatment (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings towards the treatment. The result presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction.
  scores on scale | 28.86 (6.35) | 28.62 (6.45) | 27.54 (6.55) | 28.34 (6.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Estimated mean change from baseline in HbA1c at week 30. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using mixed model for repeated measurements.
Time Frame: Week 0, week 30
Population: Full analysis set included all randomised subjects who had received at least 1 dose of randomised semaglutide or placebo.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
percentage of glycosylated hemoglobin | -1.45 (0.09) | -1.85 (0.09) | -0.09 (0.09)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Hierarchical testing was performed as per sequence listed below:Change in HbA1c: semaglutide 1.0 mg vs placebo. Change in HbA1c: semaglutide 0.5 mg vs placebo. Change in body weight: semaglutide 1.0 mg vs placebo. Change in body weight: semaglutide 0.5 mg vs placebo. Analysis was performed using MMRM with treatment, country and stratification variable (HbA1c at screening [≤8.0% or >8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.75, 95% CI 2-sided [-2.01 to -1.50] — Superiority for change in HbA1c was claimed if the upper limit of the 2-sided 95% CI for the estimated difference was below 0%
Statistical Analysis 2: Comparison: Semaglutide 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.35, 95% CI 2-sided [-1.61 to -1.10] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Body Weight
Description: Estimated mean change from baseline in body weight at week 30. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using mixed model for repeated measurements.
Time Frame: Week 0, week 30
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
kg | -3.67 (0.36) | -6.42 (0.36) | -1.36 (0.37)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Estimated mean change from baseline in FPG at week 30. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using mixed model for repeated measurements.
Time Frame: week 0, week 30
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
mg/dL | -29.14 (3.74) | -42.38 (3.76) | -8.51 (4.02)

4. Secondary Outcome: Change in Insulin Dose
Description: Estimated mean change from baseline in insulin dose at week 30 was measured in terms of ratio to baseline. Responses at week 30 are analysed using an Analysis of covariance model with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using last observation carried forward.
Time Frame: week 0, week 30
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
ratio | 0.90 (0.01) | 0.85 (0.01) | 0.96 (0.01)

5. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Estimated mean change from baseline in systolic and diastolic blood pressure at week 30. The post-baseline responses are analysed using a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using mixed model for repeated measurements.
Time Frame: week 0, week 30
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
mm Hg
  Diastolic blood pressure | -1.84 (0.73) | -1.50 (0.74) | -2.17 (0.79)
  Systolic blood pressure | -4.29 (1.26) | -7.27 (1.27) | -0.99 (1.34)

6. Secondary Outcome: Patient Reported Outcomes, Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Description: The DTSQs questionnaire was used to assess subjects' treatment satisfaction and contained 8 components and evaluates the diabetes treatment (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings towards the treatment. The result presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction. The post-baseline responses are analysed using an ANCOVA model with treatment, country and stratification variables (HbA1c level at screening [<= 8.0% or > 8.0%] and use of metformin [yes or no]) as fixed factors and baseline value as covariate. Mean estimates are adjusted according to observed baseline distribution. Missing data was imputed using last observation carried forward.
Time Frame: week 0, week 30
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
scores on a scale | 2.73 (0.46) | 3.47 (0.46) | 1.25 (0.50)

7. Secondary Outcome: HbA1c Below 7.0% (53 mmol/Mol) American Diabetes Association (ADA) Target
Description: Percentage of subjects with HbA1C below 7.0% after 30 weeks treatment. Missing data imputed from a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 30 weeks treatment
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
percentage of subjects | 60.6 | 78.6 | 10.5

8. Secondary Outcome: HbA1c Below or Equal to 6.5% (48 mmol/Mol) American Association of Clinical Endocrinologists (AACE) Target
Description: Percentage of participants with HbA1c below or equal to 6.5% after 30 weeks treatment. Missing data imputed from a mixed model for repeated measurements with treatment, country and stratification variable (HbA1c level at screening [<= 8.0% or > 8.0%] crossed with use of metformin [yes or no]; 2 by 2 levels) as fixed factors and baseline value as covariate, all nested within visit.
Time Frame: After 30 weeks treatment
Population: Full analysis set.
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 132 | 131 | 133
percentage of subjects | 40.9 | 61.1 | 4.5

ADVERSE EVENTS:
Time Frame: From the first dose of trial product until the end of the post-treatment follow-up period.The follow-up visit was scheduled to take place 5 weeks after the date of last dose of trial product with a visit window of +7 days (maximum 36 weeks).
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that had onset date (or increased in severity) during the 'on-treatment' observation period.
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/132 | 12/131 | 9/133
Other Adverse Events (participants affected / at risk) | 52/132 | 54/131 | 34/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=132) | Semaglutide 1.0 mg (N=131) | Placebo (N=133)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=132) | Semaglutide 1.0 mg (N=131) | Placebo (N=133)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 2 (2)
Lipase increased (Investigations) | 12 (15) | 7 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (14) | 6 (6) | 14 (16)
Nausea (Gastrointestinal disorders) | 15 (21) | 22 (23) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (5) | 8 (11)
Vomiting (Gastrointestinal disorders) | 8 (9) | 15 (17) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.